CLINICAL TRIAL: NCT03586362
Title: Vancomycin De-escalation Therapy in Patients With Pneumonia and Negative MRSA Nasal Swab
Brief Title: Vancomycin De-escalation Therapy in Patients With Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Rayan Ihle, M.D, CAMC Health System
Other Study IDs: 17-406
Record Dates: First submitted 2018-07-03; First posted 2018-07-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Pneumonia
Keywords: Vancomycin; MRSA nasal swab; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment Group A: Patients admitted for pneumonia whose MRSA nasal swab is negative for MRSA, and empiric vancomycin is discontinued within 24 hours of the MRSA nasal swab results being documented in the electronic health record.
- Treatment Group B: Patients admitted for pneumonia whose empiric vancomycin is continued for ≥24 hours after electronic health record documentation of negative MRSA nasal swab results.

SUMMARY:
This is a non-inferiority study evaluating clinical improvement rate when using MRSA nasal swabs to guide discontinuation of vancomycin for empiric coverage for MRSA pneumonia.

DETAILED DESCRIPTION:
Current clinical guidelines recommend including vancomycin in initial empiric therapy if risk factors for MRSA infection are present, or there is a high incidence of MRSA locally. Prolonged exposure to vancomycin, however, has been linked with the risk of vancomycin-associated kidney failure. Studies have reported that a MRSA nasal swab may be used to predict the presence of MRSA pneumonia. Specifically, pneumonia patients with negative MRSA nasal swabs are 95-99% likely to not have pneumonia due to MRSA. There is limited data, however, evaluating the use of a MRSA nasal swab to guide vancomycin therapy. Accordingly, in this study, pneumonia patients in the intervention arm will have empiric vancomycin discontinued following a negative MRSA nasal swab. In the control arm, patients vancomycin will not be discontinued based on the MRSA nasal swab result. The rate of clinical resolution will be compared between these two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Patients admitted to Charleston Area Medical Center (CAMC) through the Emergency Department who meet the CDC criteria for pneumonia.
* Nasal surveillance culture for MRSA obtained in the Emergency Department
* Patients receiving vancomycin and additional antibiotic therapy for gram-negative coverage

Exclusion Criteria:

* Persistent vasopressor requirements when MRSA nasal swab results are available
* Patients not meeting the CDC criteria for pneumonia
* Patients presenting to the ED with leukopenia (≤4000) without previous documentation of normal or elevated WBC
* Patients receiving empiric MRSA antibiotic therapy other than vancomycin for pneumonia
* Patients with the diagnosis of lung abscess
* Patients not receiving vancomycin therapy before MRSA nasal swab results are reported
* Immunocompromised individuals. i.e. patients with AIDS/HIV, vasculitis on immune suppressor therapy, steroid therapy for more than one week prior admission or who received chemotherapy in the last 3 months
* Patients who do not have a MRSA nasal swab obtained in the ED
* Nares swab obtained after the completion of the first administered dose of an antibiotic with activity against MRSA
* Patients with MRSA bacteremia
* Patients with chronic tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Charleston Area Medical Center through the Emergency Department with a diagnosis of pneumonia will be evaluated for potential enrollment.
Sampling Method: Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical Improvement | Evaluation will be completed 48 hours after 7 days of antibiotic therapy for pneumonia.
  Rate of clinical improvement following 7 days of antibiotic therapy for pneumonia. Clinical improvement rate is defined as the percentage of patients who had clinical documentation of improvement or resolution of all clinical signs and symptoms of pneumonia present at the time of pneumonia diagnosis.
  * Afebrile: Temperature <38.0ºC or <100.4ºF
  * Improvement of respiratory symptoms and signs per clinical documentation: cough, dyspnea, tachypnea, purulent sputum, increase respiratory secretions, increased suctioning requirements
  * White blood count (WBC) trending down by at least 25%, or when baseline was≤ 15,000 mm3, or return to the normal values
  * Less oxygen supplementation and ventilation
  * Chest radiographic improvement per radiologist report (e.g. infiltrate, consolidation or cavitation)

SECONDARY OUTCOMES:
Hospital Length of Stay | During patient hospital stay for up to 6 months
  Date of admission to date of discharge from the hospital
In-hospital mortality | During patient hospital stay for up to 6 months
  Number of deaths
Rate of vancomycin-associated kidney injury defined as a 50% increase in serum creatinine or at least two consecutive increases in serum creatinine by 0.5 mg/dL after at least 48 hours of vancomycin therapy. | Time between vancomycin administration and discharge from hospital for up to 6 months.
  Number of kidney injuries following administration of vancomycin
Hospital complications, such as MRSA bacteremia and septic shock | During patient hospital stay for up tp 6 months
  Number of MRSA bacteremia and septic shock patients whose MRSA nasal swab is negative and have MRSA pneumonia
Billing cost associated with vancomycin therapy and laboratory monitoring | During patient hospital stay for up to 6 months
  Total charges associated with vancomycin therapy and laboratory monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Audis Bethea, PharmD, BCPS, Principal Investigator — CAMC Health System
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States

REFERENCES:
- [Background] Edwards JR, Peterson KD, Andrus ML, Dudeck MA, Pollock DA, Horan TC; National Healthcare Safety Network Facilities. National Healthcare Safety Network (NHSN) Report, data summary for 2006 through 2007, issued November 2008. Am J Infect Control. 2008 Nov;36(9):609-26. doi: 10.1016/j.ajic.2008.08.001. No abstract available. PMID 18992647
- [Background] Greenaway CA, Embil J, Orr PH, McLeod J, Dyck B, Nicolle LE. Nosocomial pneumonia on general medical and surgical wards in a tertiary-care hospital. Infect Control Hosp Epidemiol. 1997 Nov;18(11):749-56. doi: 10.1086/647529. PMID 9397368
- [Background] Cook DJ, Kollef MH. Risk factors for ICU-acquired pneumonia. JAMA. 1998 May 27;279(20):1605-6. doi: 10.1001/jama.279.20.1605. No abstract available. PMID 9613899
- [Background] Craven DE, Steger KA. Epidemiology of nosocomial pneumonia. New perspectives on an old disease. Chest. 1995 Aug;108(2 Suppl):1S-16S. doi: 10.1378/chest.108.2_supplement.1s. No abstract available. PMID 7634921
- [Background] Zimlichman E, Henderson D, Tamir O, Franz C, Song P, Yamin CK, Keohane C, Denham CR, Bates DW. Health care-associated infections: a meta-analysis of costs and financial impact on the US health care system. JAMA Intern Med. 2013 Dec 9-23;173(22):2039-46. doi: 10.1001/jamainternmed.2013.9763. PMID 23999949
- [Background] Rubinstein E, Kollef MH, Nathwani D. Pneumonia caused by methicillin-resistant Staphylococcus aureus. Clin Infect Dis. 2008 Jun 1;46 Suppl 5:S378-85. doi: 10.1086/533594. PMID 18462093
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF; Infectious Diseases Society of America. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis. 2011 Feb 1;52(3):e18-55. doi: 10.1093/cid/ciq146. Epub 2011 Jan 4. PMID 21208910
- [Background] Erb CT, Patel B, Orr JE, Bice T, Richards JB, Metersky ML, Wilson KC, Thomson CC. Management of Adults with Hospital-acquired and Ventilator-associated Pneumonia. Ann Am Thorac Soc. 2016 Dec;13(12):2258-2260. doi: 10.1513/AnnalsATS.201608-641CME. No abstract available. PMID 27925784
- [Background] van Hal SJ, Paterson DL, Lodise TP. Systematic review and meta-analysis of vancomycin-induced nephrotoxicity associated with dosing schedules that maintain troughs between 15 and 20 milligrams per liter. Antimicrob Agents Chemother. 2013 Feb;57(2):734-44. doi: 10.1128/AAC.01568-12. Epub 2012 Nov 19. PMID 23165462
- [Background] Harigaya Y, Bulitta JB, Forrest A, Sakoulas G, Lesse AJ, Mylotte JM, Tsuji BT. Pharmacodynamics of vancomycin at simulated epithelial lining fluid concentrations against methicillin-resistant Staphylococcus aureus (MRSA): implications for dosing in MRSA pneumonia. Antimicrob Agents Chemother. 2009 Sep;53(9):3894-901. doi: 10.1128/AAC.01585-08. Epub 2009 Jul 13. PMID 19596879
- [Background] Rybak M, Lomaestro B, Rotschafer JC, Moellering R Jr, Craig W, Billeter M, Dalovisio JR, Levine DP. Therapeutic monitoring of vancomycin in adult patients: a consensus review of the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2009 Jan 1;66(1):82-98. doi: 10.2146/ajhp080434. No abstract available. PMID 19106348
- [Background] Minejima E, Choi J, Beringer P, Lou M, Tse E, Wong-Beringer A. Applying new diagnostic criteria for acute kidney injury to facilitate early identification of nephrotoxicity in vancomycin-treated patients. Antimicrob Agents Chemother. 2011 Jul;55(7):3278-83. doi: 10.1128/AAC.00173-11. Epub 2011 May 16. PMID 21576448
- [Background] Hazlewood KA, Brouse SD, Pitcher WD, Hall RG. Vancomycin-associated nephrotoxicity: grave concern or death by character assassination? Am J Med. 2010 Feb;123(2):182.e1-7. doi: 10.1016/j.amjmed.2009.05.031. PMID 20103028
- [Background] Hiramatsu K, Hanaki H, Ino T, Yabuta K, Oguri T, Tenover FC. Methicillin-resistant Staphylococcus aureus clinical strain with reduced vancomycin susceptibility. J Antimicrob Chemother. 1997 Jul;40(1):135-6. doi: 10.1093/jac/40.1.135. No abstract available. PMID 9249217
- [Background] Pitz AM, Yu F, Hermsen ED, Rupp ME, Fey PD, Olsen KM. Vancomycin susceptibility trends and prevalence of heterogeneous vancomycin-intermediate Staphylococcus aureus in clinical methicillin-resistant S. aureus isolates. J Clin Microbiol. 2011 Jan;49(1):269-74. doi: 10.1128/JCM.00914-10. Epub 2010 Oct 20. PMID 20962147
- [Background] Richter SS, Satola SW, Crispell EK, Heilmann KP, Dohrn CL, Riahi F, Costello AJ, Diekema DJ, Doern GV. Detection of Staphylococcus aureus isolates with heterogeneous intermediate-level resistance to vancomycin in the United States. J Clin Microbiol. 2011 Dec;49(12):4203-7. doi: 10.1128/JCM.01152-11. Epub 2011 Oct 5. PMID 21976769
- [Background] Tilahun B, Faust AC, McCorstin P, Ortegon A. Nasal colonization and lower respiratory tract infections with methicillin-resistant Staphylococcus aureus. Am J Crit Care. 2015 Jan;24(1):8-12. doi: 10.4037/ajcc2015102. PMID 25554549
- [Background] Hiett J, Patel RK, Tate V, Smulian G, Kelly A. Using active methicillin-resistant Staphylococcus aureus surveillance nasal swabs to predict clinical respiratory culture results. Am J Health Syst Pharm. 2015 Jun 1;72(11 Suppl 1):S20-4. doi: 10.2146/ajhp140820. PMID 25991589
- [Background] Pugin J, Auckenthaler R, Mili N, Janssens JP, Lew PD, Suter PM. Diagnosis of ventilator-associated pneumonia by bacteriologic analysis of bronchoscopic and nonbronchoscopic "blind" bronchoalveolar lavage fluid. Am Rev Respir Dis. 1991 May;143(5 Pt 1):1121-9. doi: 10.1164/ajrccm/143.5_Pt_1.1121. PMID 2024824
- [Background] Schurink CAM, Nieuwenhoven CAV, Jacobs JA, Rozenberg-Arska M, Joore HCA, Buskens E, Hoepelman AIM, Bonten MJM. Clinical pulmonary infection score for ventilator-associated pneumonia: accuracy and inter-observer variability. Intensive Care Med. 2004 Feb;30(2):217-224. doi: 10.1007/s00134-003-2018-2. Epub 2003 Oct 18. PMID 14566455
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Stevens V, Yoo, M, Brown J. Cost and Length of Stay Associated with Vancomycin-Induced Nephrotoxicity. Value in Health , Volume 16 , Issue 7 , A349
- See also: Pneumonia." Centers for Disease Control and Prevention. Centers for Disease Control and Prevention, 06 Oct. 2016. Web. 18 Jan. 2017 — https://www.cdc.gov/nchs/fastats/pneumonia.htm
- See also: 19. Centers for Disease Control and Prevention. Centers for Disease Control and Prevention, n.d. Web. 26 Jan. 2017 — https://www.cdc.gov/mmwr/preview/mmwrhtml/mm5126a1.htm